CLINICAL TRIAL: NCT03381729
Title: Phase I, Open-Label, Dose Comparison Study of AVXS-101 for Sitting But Non-ambulatory Patients With Spinal Muscular Atrophy
Brief Title: Study of Intrathecal Administration of Onasemnogene Abeparvovec-xioi for Spinal Muscular Atrophy
Acronym: STRONG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based upon overall strategic objectives within the broader intrathecal clinical development program, Novartis Gene Therapies decided to terminate the study early.
Sponsor: Novartis Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVXS-101-CL-102; 2020-003678-28 (EudraCT Number); COAV101A12102 (Other: Novartis)
Record Dates: First submitted 2017-12-13; First posted 2017-12-22 (Actual); Results first posted 2023-02-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy
Keywords: Gene Transfer; Gene Therapy; Adeno-associated virus; Survival Motor Neuron; SMN; AAV9
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Zolgensma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose A (Experimental): Intrathecal administration 6.0 X 10^13 vg of onasemnogene abeparvovec-xioi
  Interventions: Biological: Onasemnogene Abeparvovec-xioi
- Dose B (Experimental): Intrathecal administration 1.2 X 10^14 vg of onasemnogene abeparvovec-xioi
  Interventions: Biological: Onasemnogene Abeparvovec-xioi
- Dose C (Experimental): Intrathecal administration 2.4 X 10^14 vg of onasemnogene abeparvovec-xioi
  Interventions: Biological: Onasemnogene Abeparvovec-xioi

INTERVENTIONS:
Biological: Onasemnogene Abeparvovec-xioi — Self-complementary AAV9 carrying the SMN gene under the control of a hybrid CMV enhancer/chicken-β-actin promoter
  Other Names: Zolgensma

SUMMARY:
The purpose of this trial is to evaluate the safety and tolerability of intrathecal administration of onasemnogene abeparvovec-xioi in infants and children with Spinal Muscular Atrophy with 3 copies of SMN2 and deletion of SMN1.

DETAILED DESCRIPTION:
This is a Phase 1, single-dose administration study of infants and children with a genetic diagnosis consistent with spinal muscular atrophy (SMA), bi-allelic deletion of survival motor neuron 1 gene (SMN1) and 3 copies of survival motor neuron 2 gene (SMN2) without the genetic modifier who are able to sit but cannot stand or walk at the time of study entry. Patients will receive onasemnogene abeparvovec-xioi in a dose comparison safety study of two (or three) potential therapeutic doses. Patients will be stratified in two groups, those ≥6 months and < 24 months of age at time of dosing and those ≥ 24 months and < 60 months of age at time of dosing. At least 15 patients ≥ 6 months and < 24 months, and at least 12 patients ≥ 24 < 60 months will be enrolled.

The first cohort will enroll three patients (Cohort 1) ≥ 6 months and < 24 months of age who will receive administration of 6.0 × 1013 vg of onasemnogene abeparvovec-xioi (Dose A). There will be at least a four week interval between the dosing of each patient within the cohort. Novartis Gene Therapies, Inc. will confer with the Data Safety Monitoring Board (DSMB) on all Grade III or higher AEs within approximately 48 hours of awareness that are possibly, probably or definitely related to the study agent before continuing enrollment. Safety data will be reviewed by the DSMB during quarterly meetings; following enrollment of the three patients and based upon the available safety data a decision will be made whether to: a) stop due to toxicity, or b) proceed to Cohort 2 using Dose B.

Should the determination be made to advance to Dose B, three patients < 60 months of age will be enrolled (Cohort 2) and will receive administration of 1.2 × 1014 vg of onasemnogene abeparvovec-xioi (Dose B). Again, there will be at least a four-week interval between dosing of the three patients within the cohort. Based on the available safety data from the three Cohort 2 patients and all of the Cohort 1 patients, the DSMB will decide and document during quarterly meetings whether further four-week intervals between patients dosing is necessary. Novartis Gene Therapies, Inc. will take this recommendation into consideration and will make the final determination whether to persist with four-week intervals between patients dosing going forward; the decision will be communicated to sites and Institutional Review Boards (IRBs) in a formal sponsor letter. Novartis Gene Therapies, Inc. will confer with the DSMB on all Grade III or higher AEs within approximately 48 hours of awareness that are possibly, probably or definitely related to the study agent before continuing enrollment. Safety data will be reviewed by the DSMB during quarterly meetings; following enrollment of the first six patients and based upon available safety data, a decision will be made whether to: a) stop due to toxicity, or b) continue to enroll an additional 21 patients until there are a total of 12 patients > 6 months and < 24 months and 12 patients ≥ 24 and < 60 months that have all received Dose B.

Based upon an ongoing assessment of safety and efficacy data from patients treated with the 1.2 × 1014 vg dose, an option for testing of a third dose (Dose C), will be considered. If, based on all available data, this is judged to be safe and necessary, three patients < 60 months of age will receive Dose C, 2.4 × 1014 vg administered IT. A meeting of the DSMB will be called to obtain a recommendation on the safety of escalating to a higher dose prior to proceeding. If a decision is made to proceed to testing a higher dose, there will again be a four-week interval between dosing of the first three patients receiving Dose C, as in Cohorts 1 and 2. Safety data will be reviewed by the DSMB during quarterly meetings. Following enrollment of the first three Dose C patients and based upon available safety data, the DSMB will be consulted and a decision will be made whether to: a) stop dosing Dose C due to safety concerns, or b) continue to enroll an additional 21 patients until there are a total of 12 patients > 6 months and < 24 months and 12 patients ≥ 24 and < 60 months that have received Dose C.

Patients from Cohort 3 will be followed for a total of 15 months post-dose. The primary analyses for efficacy will be assessed when all patients reach 12 months post-dose and the primary analyses for safety will be assessed when the last patient of Cohort 3 reaches 15 months post-dose (and database lock will be performed after the last patient reaches 15 months post-dose).

ELIGIBILITY:
Key Inclusion Criteria

* Patients ≥6 months and up to 60 months (1800 days) of age at time of dosing following diagnostic confirmation during screening period by genotype who demonstrate the ability to sit unassisted for 10 or more seconds but cannot stand or walk
* Diagnostic confirmation by genotype includes lab documentation of homozygous absence of SMN1 exon 7; with exactly three copies of SMN2
* Negative gene testing for SMN2 gene modifier mutation (c.859G>C)
* Onset of clinical signs and symptoms consistent with spinal muscular atrophy (SMA) at < 12 months of age
* Able to sit independently and not standing or walking independently. Definition of sitting independently is defined by the World Health Organization Multicentre Growth Reference Study (WHO-MGRS) criteria of being able to sit up unsupported with head erect for at least 10 seconds. Child should not use arms or hands to balance body or support position (Wijnhoven 2004)
* Be up-to-date on childhood vaccines that include palivizumab prophylaxis (also known as Synagis) to prevent respiratory syncytial virus (RSV) infections are also recommended in accordance with American Academy of Pediatrics (AAP 2009)

Key Exclusion Criteria

* Current or historical ability to stand or walk independently
* Contraindications for spinal tap procedure or administration of intrathecal therapy or presence of an implanted shunt for the drainage of CSF or an implanted central venous (CNS) catheter
* Severe contractures as determined by designated Physical Therapist(s) at screening that interfere with either the ability to attain/demonstrate functional measures or interferes with ability to receive intrathecal (IT) dosing
* Severe scoliosis (defined as ≥ 50° curvature of spine) evident on X-ray examination
* Previous, planned or expected scoliosis repair surgery/procedure within 1 year of dose administration
* Use of invasive ventilatory support (tracheotomy with positive pressure) or pulse oximetry < 95% saturation at screening while the patient is awake, or for high altitudes > 1000 m, oxygen saturation < 92% while the patient is awake
* Pulse oximetry saturation must not decrease ≥ four (4) percentage points between screening and highest value on day of dosing
* Use or requirement of non-invasive ventilatory support for 12 or more hours daily over the two (2) weeks prior to dosing
* Medical necessity for a gastric feeding tube, where the majority of feedings are given by non-oral methods (i.e., nasogastric tube or nasojejunal tube) or patients whose weight-for-age falls below the 3rd percentile based on WHO Child Growth Standards (Onis 2006). Placement of a permanent gastrostomy prior to screening is not an exclusion
* Use or requirement of non-invasive ventilatory support for 12 or more hours daily over the two (2) weeks prior to dosing
* Medical necessity for a gastric feeding tube, where the majority of feedings are given by non-oral methods or patients whose weight-for-age falls below the 3rd percentile based on WHO Child Growth Standards (Onis 2006). Placement of a permanent gastrostomy prior to screening is not an exclusion
* Active viral infection (includes human immunodeficiency virus (HIV) or serology positive for hepatitis B or C, or Zika virus)
* Serious non-respiratory tract illness requiring systemic treatment and/or hospitalization within two (2) weeks prior to study entry
* Respiratory infection requiring medical attention, medical intervention or increase in supportive care of any manner within four (4) weeks prior to study entry
* Severe non-pulmonary/respiratory tract infection within four (4) weeks before study dosing or concomitant illness that in the opinion of the Principal Investigator (PI) creates unnecessary risks for gene transfer such as:

  * Major renal or hepatic impairment
  * Known seizure disorder
  * Diabetes mellitus
  * Idiopathic hypocalciuria
  * Symptomatic cardiomyopathy
* History of bacterial meningitis or brain or spinal cord disease, including tumors, or abnormalities by magnetic resonance imaging (MRI) or computerized tomography (CT) that would interfere with the lumbar puncture (LP) procedures or CSF circulation
* Known allergy or hypersensitivity to prednisolone or other glucocorticosteroids or their excipients
* Known allergy or hypersensitivity to iodine or iodine-containing products
* Concomitant use of any of the following: drugs for treatment of myopathy or neuropathy, agents used to treat diabetes mellitus, or ongoing immunosuppressive therapy, plasmapheresis, immunomodulators such as adalimumab, or immunosuppressive therapy within 3 months of study dosing
* Inability to withhold use of laxatives or diuretics in the 24 hours prior to dose administration
* Anti-AAV9 antibody titers >1:50 as determined by Enzyme-linked Immunosorbent Assay (ELISA) binding immunoassay

  * Should a potential patient demonstrate anti AAV9 antibody titer > 1:50, he or she may receive retesting within 30 days of the screening period and will be eligible to participate if the anti AAV9 antibody titer upon retesting is ≤ 1:50
* Clinically significant abnormal laboratory values (GGT, ALT, and AST, or total bilirubin > 2 × ULN, creatinine ≥ 1.0 mg/dL, hemoglobin [Hgb] < 8 or > 18 g/dL; white blood cell [WBC] > 20,000 per cmm) prior to gene replacement therapy. Patients with an elevated bilirubin level that is unequivocally the result of neonatal jaundice shall not be excluded
* Participation in recent SMA treatment clinical trial or receipt of an investigational or approved compound product or therapy received with the intent to treat SMA at any time prior to screening for this study

  * Oral beta agonists must be discontinued 30 days prior to dosing.
  * Inhaled albuterol specifically prescribed for the purposes of respiratory (bronchodilator) management is acceptable and not a contraindication at any time prior to screening for this study
* Expectation of major surgical procedures during the 1-year study assessment period

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - Nemours Children's Hospital, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Duque SI, Arnold WD, Odermatt P, Li X, Porensky PN, Schmelzer L, Meyer K, Kolb SJ, Schumperli D, Kaspar BK, Burghes AH. A large animal model of spinal muscular atrophy and correction of phenotype. Ann Neurol. 2015 Mar;77(3):399-414. doi: 10.1002/ana.24332. Epub 2015 Feb 9. PMID 25516063
- [Background] Foust KD, Wang X, McGovern VL, Braun L, Bevan AK, Haidet AM, Le TT, Morales PR, Rich MM, Burghes AH, Kaspar BK. Rescue of the spinal muscular atrophy phenotype in a mouse model by early postnatal delivery of SMN. Nat Biotechnol. 2010 Mar;28(3):271-4. doi: 10.1038/nbt.1610. Epub 2010 Feb 28. PMID 20190738 (Retraction: PMID 36203015 Nat Biotechnol. 2022 Nov;40(11):1692)
- [Background] Meyer K, Ferraiuolo L, Schmelzer L, Braun L, McGovern V, Likhite S, Michels O, Govoni A, Fitzgerald J, Morales P, Foust KD, Mendell JR, Burghes AH, Kaspar BK. Improving single injection CSF delivery of AAV9-mediated gene therapy for SMA: a dose-response study in mice and nonhuman primates. Mol Ther. 2015 Mar;23(3):477-87. doi: 10.1038/mt.2014.210. Epub 2014 Oct 31. PMID 25358252
- See also: The Novartis Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17933
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1220

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 participants took part in the trial at 11 sites in the United States between December 2017 and May 2021.
Pre-assignment Details: A total of 38 participants were screened, of which 6 were screen failures and 32 were enrolled and received study drug.
Groups:
- Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months: Participants aged 6 to <24 months at time of AVXS-101 dosing received a single 6.0E13 vg dose of AVXS-101 administered as an intrathecal injection on Day 1 of the overall study. Participants also received daily doses of prophylactic oral prednisolone starting at a dose of 1 mg/kg/day from 1 day prior to AVXS-101 injection until at least 30 days post-injection at which point the prednisolone dose could be tapered downwards. At week 9, prednisolone could be discontinued.
- Cohort 2: 1.2E14 vg - Age 6 to <24 Months: Participants aged 6 to <24 months at time of AVXS-101 dosing received a single 1.2E14 vg dose of AVXS-101 administered as an intrathecal injection on Day 1 of the overall study. Participants also received daily doses of prophylactic oral prednisolone starting at a dose of 1 mg/kg/day from 1 day prior to AVXS-101 injection until at least 30 days post-injection at which point the prednisolone dose could be tapered downwards. At week 9, prednisolone could be discontinued.
- Cohort 2: 1.2E14 vg - Age 24 to <60 Months: Participants aged 24 to <60 months at time of AVXS-101 dosing received a single 1.2E14 vg dose of AVXS-101 administered as an intrathecal injection on Day 1 of the overall study. Participants also received daily doses of prophylactic oral prednisolone starting at a dose of 1 mg/kg/day from 1 day prior to AVXS-101 injection until at least 30 days post-injection at which point the prednisolone dose could be tapered downwards. At week 9, prednisolone could be discontinued.
- Cohort 3: 2.4E14 vg - Age 6 to <24 Months: Participants aged 6 to <24 months at time of AVXS-101 dosing received a single 2.4E14 vg dose of AVXS-101 administered as an intrathecal injection on Day 1 of the overall study. Participants also received daily doses of prophylactic oral prednisolone starting at a dose of 1 mg/kg/day from 1 day prior to AVXS-101 injection until at least 30 days post-injection at which point the prednisolone dose could be tapered downwards. At week 9, prednisolone could be discontinued.
- Cohort 3: 2.4E14 vg - Age 24 to <60 Months: Participants aged 24 to <60 months at time of AVXS-101 dosing were planned to receive a single 2.4E14 vg dose of AVXS-101 administered as an intrathecal injection on Day 1 of the overall study. Participants were also planned to receive daily doses of prophylactic oral prednisolone starting at a dose of 1 mg/kg/day from 1 day prior to AVXS-101 injection until at least 30 days post-injection at which point the prednisolone dose could have been tapered downwards. At week 9, prednisolone could have been discontinued. Due to early termination of the study, no participants aged 24 to <60 months were enrolled in Cohort 3.
Period: Overall Study
Arm/Group | Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 24 to <60 Months | Cohort 3: 2.4E14 vg - Age 6 to <24 Months | Cohort 3: 2.4E14 vg - Age 24 to <60 Months
Started | 3 | 13 | 12 | 4 | 0
Received AVXS-101 | 3 | 13 | 12 | 4 | 0
Completed | 3 | 13 | 12 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants given an AVXS-101 intrathecal injection. Participants were analyzed according to actual dose received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 24 to <60 Months | Cohort 3: 2.4E14 vg - Age 6 to <24 Months | Total
Number analyzed (Participants) | 3 | 13 | 12 | 4 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 13 | 12 | 4 | 32
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 17.2 (4.1) | 16.7 (4.5) | 37.5 (10.6) | 16.9 (5.6) | 24.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 6 | 0 | 14
  Male | 1 | 7 | 6 | 4 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 0 | 5
  Not Hispanic or Latino | 1 | 10 | 12 | 4 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 10 | 8 | 3 | 23
  Asian | 0 | 1 | 4 | 1 | 6
  Other | 0 | 1 | 0 | 0 | 1
  Multiple | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Age 6 to <24 Months Only: Number of Participants Who Achieved the Ability to Stand Alone
Description: Defined by the Bayley Scales of Infant and Toddler Development (BSID) Gross Motor (GM) subtest performance criteria number 40, confirmed by video recording, as a participant who stands alone for at least 3 seconds unsupported.
Time Frame: From Day 1 up to Month 12
Population: Intent-to-Treat (ITT) Set: All enrolled participants who were given an AVXS-101 intrathecal injection. Participants were analyzed according to the assigned dose. Data were only collected in participants aged 6 to <24 months at time of dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 6 to <24 Months | Cohort 3: 2.4E14 vg - Age 6 to <24 Months
Number analyzed (Participants) | 3 | 13 | 4
Participants
  Able to Stand Alone | 1 | 1 | 0
  Unable to Stand Alone | 2 | 12 | 4
Statistical Analysis 1: Comparison: Cohort 2: 1.2E14 vg - Age 6 to <24 Months; Difference in the percentage of participants who achieved the ability to stand alone; Test type: Superiority; p > 0.9999, Fisher Exact; Difference in Percent = -6.0, 95% CI 2-sided [-21.8 to 22.8]; Data for the current study were compared to historical control data (Finkel et al 2014 - PubMed 25080519) where 7 (13.7%) participants achieved the ability to stand alone and 44 (86.3%) participants did not achieve the ability to stand alone

2. Primary Outcome: Age 24 to <60 Months Only: Change From Baseline in Hammersmith Functional Motor Scale-Expanded (HFMSE) Score at Month 12
Description: The HFMSE contained 33 items which were scored on a scale of 0-2 with a total achievable score ranging from 0, if all activities are failed, to 66, if all the activities are achieved. A positive change from baseline indicates a better outcome.
Time Frame: Baseline and Month 12
Population: ITT Set: All enrolled participants who were given an AVXS-101 intrathecal injection. Participants were analyzed according to the assigned dose. Data were only collected in participants aged 24 to <60 months at time of dosing.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cohort 2: 1.2E14 vg - Age 24 to <60 Months
Number analyzed (Participants) | 12
score on a scale | 6.0 [3.7 to 8.3]
Statistical Analysis 1: Comparison: Cohort 2: 1.2E14 vg - Age 24 to <60 Months; Test type: Superiority; p = 0.0027, Mixed-Model Repeat Measure; Difference Between Least Squares Mean = 5.5, 95% CI 2-sided [1.9 to 9.0]; Data for the current study were compared to historical control data (Finkel et al 2014 - PubMed 25080519) where the least squares mean (95% confidence interval) of the change from baseline in HFMSE scores at 12 months was 0.5 (-2.2 to 3.2)

3. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any event that began or worsened in severity on or after the administration of AVXS-101 through the last study visit.
  Evaluation of TEAEs included the number of participants with at least one:
  * TEAE
  * Serious TEAE
  * TEAE related to AVXS-101
  * TEAE with Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 (grade 3 = severe or medically significant to grade 5 = death related to TEAE)
Time Frame: Adverse events were collected from the single dose of study treatment until the end of study visit (12 months for Cohort 1 and 2 and 15 months for Cohort 3)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 24 to <60 Months | Cohort 3: 2.4E14 vg - Age 6 to <24 Months
Number analyzed (Participants) | 3 | 13 | 12 | 4
Participants
  TEAE | 3 | 13 | 12 | 4
  Serious TEAE | 1 | 2 | 4 | 0
  TEAE Related to AVXS-101 | 0 | 7 | 4 | 1
  TEAE with CTCAE Grade ≥ 3 | 1 | 4 | 4 | 0

4. Secondary Outcome: Number of Participants Who Achieved the Ability to Walk Alone
Description: Defined by the BSID GM subtest performance criteria number 43, confirmed by video recording, as a participant who takes 5 coordinated independent steps.
Time Frame: From Day 1 up to Month 12
Population: ITT Set: All enrolled participants who were given an AVXS-101 intrathecal injection. Participants were analyzed according to the assigned dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 24 to <60 Months | Cohort 3: 2.4E14 vg - Age 6 to <24 Months
Number analyzed (Participants) | 3 | 13 | 12 | 4
Participants
  Able to Walk Alone | 0 | 1 | 0 | 0
  Unable to Walk Alone | 3 | 12 | 12 | 4
Statistical Analysis 1: Comparison: Cohort 2: 1.2E14 vg - Age 6 to <24 Months; Difference in the percentage of participants who achieved the ability to walk alone; Test type: Superiority; p > 0.9999, Fisher Exact; Percentage Difference = -2.1, 95% CI 2-sided [-17.2 to 27.0]; Data for the current study were compared to historical control data (Finkel et al 2014 PubMed 25080519) where 5 (9.8%) participants achieved the ability to walk alone and 46 (90.2%) participants did not achieve the ability to walk alone

5. Secondary Outcome: Average Number of Hours Per Day of Non-invasive Ventilatory Support
Description: Participants were assessed by a pulmonologist and may have been fitted with a non-invasive positive pressure ventilatory (e.g., Bilevel Positive Airway Pressure BiPAP) at the discretion of the pulmonologist and/or investigator. The number of hours per day of non-invasive ventilatory support was captured continuously by the device.
Time Frame: Months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
Population: Data were only collected in participants requiring BiPAP support.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 24 to <60 Months | Cohort 3: 2.4E14 vg - Age 6 to <24 Months
Number analyzed (Participants) | 0 | 1 | 1 | 0
hours/day
  Month 2: number analyzed (Participants) | 0 | 0 | 1 | 0
  Month 2 |  |  | 10.530 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 3: number analyzed (Participants) | 0 | 0 | 1 | 0
  Month 3 |  |  | 2.930 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 4 |  | 0.000 (NA) — Only 1 participant had available data so standard deviation could not be calculated. | 5.860 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 5 |  | 0.000 (NA) — Only 1 participant had available data so standard deviation could not be calculated. | 4.610 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 6 |  | 2.590 (NA) — Only 1 participant had available data so standard deviation could not be calculated. | 4.490 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 7 |  | 4.550 (NA) — Only 1 participant had available data so standard deviation could not be calculated. | 7.490 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 8 |  | 7.170 (NA) — Only 1 participant had available data so standard deviation could not be calculated. | 8.290 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 9 |  | 8.690 (NA) — Only 1 participant had available data so standard deviation could not be calculated. | 7.690 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 10 |  | 10.320 (NA) — Only 1 participant had available data so standard deviation could not be calculated. | 9.900 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 11 |  | 14.050 (NA) — Only 1 participant had available data so standard deviation could not be calculated. | 3.460 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |
  Month 12 |  | 10.120 (NA) — Only 1 participant had available data so standard deviation could not be calculated. | 0.040 (NA) — Only 1 participant had available data so standard deviation could not be calculated. |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the single dose of study treatment until the end of study visit (12 months for Cohort 1 and 2 and 15 months for Cohort 3)
Description: Safety Analysis Set: All participants given an AVXS-101 intrathecal injection. Participants were analyzed according to actual dose received.
Arm/Group | Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 6 to <24 Months | Cohort 2: 1.2E14 vg - Age 24 to <60 Months | Cohort 3: 2.4E14 vg - Age 6 to <24 Months
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/13 | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/13 | 4/12 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 13/13 | 12/12 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months (N=3) | Cohort 2: 1.2E14 vg - Age 6 to <24 Months (N=13) | Cohort 2: 1.2E14 vg - Age 24 to <60 Months (N=12) | Cohort 3: 2.4E14 vg - Age 6 to <24 Months (N=4)
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 6.0E13 Vector Genomes (vg) - Age 6 to <24 Months (N=3) | Cohort 2: 1.2E14 vg - Age 6 to <24 Months (N=13) | Cohort 2: 1.2E14 vg - Age 24 to <60 Months (N=12) | Cohort 3: 2.4E14 vg - Age 6 to <24 Months (N=4)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Pectus carinatum (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Pectus excavatum (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5 | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 2 | 3 | 2
Teething (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tooth resorption (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 6 | 7 | 2
Application site irritation (General disorders) | 0 | 1 | 0 | 0
Infusion site bruising (General disorders) | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 10 | 5 | 3
Nasopharyngitis (Infections and infestations) | 0 | 3 | 2 | 1
Otitis media (Infections and infestations) | 1 | 0 | 3 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral rash (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 1 | 0 | 0
Blood lead increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0
Carnitine decreased (Investigations) | 0 | 0 | 1 | 0
Crystal urine present (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0
Norovirus test positive (Investigations) | 0 | 0 | 0 | 1
Respirovirus test positive (Investigations) | 0 | 1 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Language disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep terror (Psychiatric disorders) | 1 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 7 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0
Aortic dilatation (Vascular disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
A comparison of the results from this study to the results from the natural history observational study (Pediatric Neuromuscular Clinical Research Network (PNCR), Finkel et al, 2014) are included in the Novartis Clinical Trial Results, as a historical control. These full results are available via this link: https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17933

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Depending on local requirements, Sponsor's consent necessary before publication of study, or Sponsor can review results communications before public release with a right to request changes to communications regarding trial results between 40 to 60 and up to 90 or 120 days, as applicable, from the time submitted to Sponsor for review to remove references to Sponsor's Confidential Information or delay results communications to permit Sponsor to obtain appropriate Intellectual Property protection.

DOCUMENTS (2):
  • Study Protocol (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03381729/Prot_002.pdf
  • Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT03381729/SAP_003.pdf